CLINICAL TRIAL: NCT04375111
Title: Comparison Between Serratus Anterior Plane Block, and Transversus Thoracic Plane Block Combined With Serratus Anterior Plane Block, for the Management of Post-mastecomy Pain.
Brief Title: Serratus Anterior Plane (SAP) Block vs SAP Block Combined With Transverus Thoracic Plane (TTP) Block, for Post-mastectomy Pain Control.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed wahby Shamsedine, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: post-mastectomy pain control
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Pain, Postoperative
Keywords: serratus anterior plane block; transversus thoracic plane block; post-mastectomy pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAP block for management of post-mastectomy pain (Active Comparator): the patients in this group shall undergo Serraturs anterior plane block for management of post-mastectomy pain.
  Interventions: Procedure: Serratus anterior plane block
- TTP block combined with SAP block for post-mastectomy pain (Active Comparator): the patients in this group shall undergo combined Serraturs anterior plane block, and Transversus thoracic plane block for management of post-mastectomy pain.
  Interventions: Procedure: Serratus anterior plane block; Procedure: Transversus thoracic plane block

INTERVENTIONS:
Procedure: Serratus anterior plane block — •Serratus anterior plane block will be carried out with the patient lying in the lateral position. After skin disinfection, the ultrasound probe will be applied parallel to and between the 5th and 6th ribs in the mid axillary region, for identification of the superficial latissimus dorsi muscles and deep anterior serratus muscles. Then, 25 ml of isobaric bupivacaine 0.25% will be injected above the serratus anterior muscle.
  Other Names: SAP block
Procedure: Transversus thoracic plane block — •Transversus thoracic plane block will be carried out with the patient lying in the supine position. After skin disinfection, the ultrasound probe will be applied parallel to and between the 4th and 5th ribs connecting at the sternum. Then, 15 ml of isobaric bupivacaine 0.25% will be injected between the transversus thoracic muscle and the internal intercosatal muscle.
  Other Names: TTP block
  Arms: TTP block combined with SAP block for post-mastectomy pain

SUMMARY:
a comparison shall be conducted between Serratus anterior plane block, on one hand, and transversus thoracic plane block combined with Serratus anterior plane block, on the other hand for management of post-mastectomy pain. VAS "Visual Analogue Scale" score will be compared in both case, and control groups.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers in women all over the world. In the united states, according to the CDC "Center of Disease Control", it's the second most common cancer occurring in women. Perioperative pain after breast surgeries remains to be taken lightly due to the minimal invasiveness of breast surgeries. However, it is estimated that 25-60% of patients undergoing breast cancer related surgeries develop chronic pain. Acute post-operative pain remains an important risk factor in developing chronic post-mastectomy pain; about 40% of women will have acute post-operative pain, on the other hand, 50% will have chronic pain. Different regional anaesthesia techniques have achieved better management of post-breast surgery acute pain and subsequently less frequent chronic pain. Add to that, effective regional anaesthesia will decrease both the surgical stress response and the requirements of general anaesthetics and opioids, which will keep the function of the immune system intact. A lot of regional anaesthesia techniques have been used to control anterior chest wall pain as the pectoral nerves (PECs) block, paravertebral block, intercostal nerve blocks, thoracic epidural analgesia, serratus anterior plane block. The breast receives its innervation through the anterior and lateral cutaneous branches of the 2nd to the 6th intercostal nerves. Targeting the serratus plane is a safer and a simpler procedure than multiple intercostal or paravertebral blocks. As a setback for the serratus anterior plane block, it only blocks the lateral cutaneous branches of the intercostal nerves with minimal if any effect on the anterior cutaneous branches. The serratus anterior plane block, being unable to block the anterior cutaneous branches of the intercostal nerves, have to be combined with another technique, transversus thoracic plane block, which can block them. The investigators here are trying to measure the efficacy of the combined serratus anterior plane block and tranversus thoracic plane block on the management of post-mastectomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients > 30 years old, ASA "American Society of Anaesthesiologists" physical status I or II undergoing any unilateral mastectomy.

Exclusion Criteria:

* Patient's refusal.
* Known contraindications to regional blocks, including local skin infections,and coagulopathy.
* Allergies to the local anaesthetics used.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Total sum of used IV additional opioid analgesia. | 24 hours post-operatively
  If the patient experiences a pain of > 3, IV morphine will be given at a dose of 2.5-5 mg per dose, with a maximum dose of 10 mg, aiming for a pain score of ≤ 3. the total morphine dose for the post-operative 24 hours will be compared between the case and control group, in order to determine which technique provided more analgesia.

SECONDARY OUTCOMES:
Post-operative pain score | 24 hours post-operatively
  VAS (Visual Analogue Scale, 0-100 mm; where 0 = no pain, and 100 = worst imaginable pain) will be assessed, at rest, per hour for 24 hours post operatively. Moreover, VAS will also be assessed at 12 and 24 hours post-operatively while abducting the ipsilateral arm. If the patient experiences a pain of > 3, IV morphine will be given at a dose of 2.5-5 mg per dose, with a maximum dose of 10 mg, aiming for a pain score of ≤ 3.

CONTACTS AND LOCATIONS:
Overall Officials: Zein El-Abdeen Z Hassan, Professor, Study Chair — Assiut University Hospitals; Montasser A Mohamed, A.Professor, Study Director — South Egypt Cancer Institute, Assiut University Hospitals.; Ahmed H Othman, A.Professor, Study Director — South Egypt Cancer Institute, Assiut University Hospitals.; Ahmed W Mohamed Shamsedine, MBBCH, Principal Investigator — South Egypt Cancer Institute, Assiut University Hospitals.
Locations (1):
- South Egypt Cancer Institute, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the decision shall be taken at the end of the study. I anticipate that it is going to be a "yes".

REFERENCES:
- [Background] DeSantis C, Ma J, Bryan L, Jemal A. Breast cancer statistics, 2013. CA Cancer J Clin. 2014 Jan-Feb;64(1):52-62. doi: 10.3322/caac.21203. Epub 2013 Oct 1. PMID 24114568
- [Background] Mejdahl MK, Andersen KG, Gartner R, Kroman N, Kehlet H. Persistent pain and sensory disturbances after treatment for breast cancer: six year nationwide follow-up study. BMJ. 2013 Apr 11;346:f1865. doi: 10.1136/bmj.f1865. PMID 23580693
- [Background] Hirko KA, Soliman AS, Hablas A, Seifeldin IA, Ramadan M, Banerjee M, Harford JB, Chamberlain RM, Merajver SD. Trends in Breast Cancer Incidence Rates by Age and Stage at Diagnosis in Gharbiah, Egypt, over 10 Years (1999-2008). J Cancer Epidemiol. 2013;2013:916394. doi: 10.1155/2013/916394. Epub 2013 Oct 24. PMID 24282410
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Lynch EP, Welch KJ, Carabuena JM, Eberlein TJ. Thoracic epidural anesthesia improves outcome after breast surgery. Ann Surg. 1995 Nov;222(5):663-9. doi: 10.1097/00000658-199511000-00009. PMID 7487214
- [Background] Kairaluoma PM, Bachmann MS, Rosenberg PH, Pere PJ. Preincisional paravertebral block reduces the prevalence of chronic pain after breast surgery. Anesth Analg. 2006 Sep;103(3):703-8. doi: 10.1213/01.ane.0000230603.92574.4e. PMID 16931684
- [Background] Huang TT, Parks DH, Lewis SR. Outpatient breast surgery under intercostal block anesthesia. Plast Reconstr Surg. 1979 Mar;63(3):299-303. doi: 10.1097/00006534-197903000-00001. PMID 419209
- [Background] Atanassoff PG, Alon E, Pasch T, Ziegler WH, Gautschi K. Intercostal nerve block for minor breast surgery. Reg Anesth. 1991 Jan-Feb;16(1):23-7. PMID 2007101
- [Background] Zocca JA, Chen GH, Puttanniah VG, Hung JC, Gulati A. Ultrasound-Guided Serratus Plane Block for Treatment of Postmastectomy Pain Syndromes in Breast Cancer Patients: A Case Series. Pain Pract. 2017 Jan;17(1):141-146. doi: 10.1111/papr.12482. Epub 2016 Sep 2. PMID 27587333
- [Background] Sarhadi NS, Shaw Dunn J, Lee FD, Soutar DS. An anatomical study of the nerve supply of the breast, including the nipple and areola. Br J Plast Surg. 1996 Apr;49(3):156-64. doi: 10.1016/s0007-1226(96)90218-0. PMID 8785595
- [Background] Mayes J, Davison E, Panahi P, Patten D, Eljelani F, Womack J, Varma M. An anatomical evaluation of the serratus anterior plane block. Anaesthesia. 2016 Sep;71(9):1064-9. doi: 10.1111/anae.13549. Epub 2016 Jul 20. PMID 27440171
- [Background] Ueshima H, Kitamura A. Blocking of Multiple Anterior Branches of Intercostal Nerves (Th2-6) Using a Transversus Thoracic Muscle Plane Block. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):388. doi: 10.1097/AAP.0000000000000245. No abstract available. PMID 26079353
- [Background] Ueshima H, Otake H. RETRACTED: Addition of transversus thoracic muscle plane block to pectoral nerves block provides more effective perioperative pain relief than pectoral nerves block alone for breast cancer surgery. Br J Anaesth. 2017 Mar 1;118(3):439-443. doi: 10.1093/bja/aew449. No abstract available. PMID 28203723 (Retraction: PMID 35219477 Br J Anaesth. 2022 Mar;128(3):598)